CLINICAL TRIAL: NCT05206617
Title: 3 Year Follow up on Patients With Pathogenic Anoctamin 5 Variants
Brief Title: 3 Year Follow up on ANO5 Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Funding: Toyota Foundation (Unknown); The Hede Nielsen Family Foundation (Other); Funding: Grosserer L. F. Foghts Foundation (Unknown); Funding: Torben og Alice Frimodts Foundation (Unknown); Funding: Aase og Ejnar Danielsens Foundation (Unknown); Funding: Oda og Hans Svenningens Foundation (Unknown); Funding: Torkild Steensbecks Legat (Unknown); Funding: Foundation for research in Neurology (Unknown)
Responsible Party: Principal Investigator, Nanna Scharff Poulsen, Principal investigator, Rigshospitalet, Denmark
Other Study IDs: H-16030358
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Neuromuscular Diseases; Limb Girdle Muscular Dystrophy
Keywords: MRI; Neuromuscular disorder; Outcome measure; Progression
MeSH Terms: conditions — Neuromuscular Diseases; Muscular Dystrophies, Limb-Girdle; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Limb Girdle Muscular Dystrophy type 2L: At baseline, 1- and 3-year follow up will the outcome measures be assessed. There will be no intervention.
  Interventions: Other: No intervention - pure observational study

INTERVENTIONS:
Other: No intervention - pure observational study — No intervention

SUMMARY:
The aim of the study is to investigate progression in muscle affection in patients with pathogenic variants in the anoctamin 5 gene to:

1. investigate possible progression of disease over time
2. investigate good and reliable outcome measures

DETAILED DESCRIPTION:
Muscles of patients with pathogenic variants in the anoctamin 5 gene will over time be infiltrated with fat. This is especially visible on MRI and can be seen even before any symptoms appear. MRI is thus used increasingly to investigate muscle affection in neuromuscular disorders. Together with functional measurements it is possible to describe how patients are affected clinically and subclinically. There are still many things that need covering - rate of progression is undertermined and good outcome measures are still needed for future clinical trials.

Muscles of the whole body in patients with neuromuscular disorders will be investigated 3 times through a 3 year follow-up study.

The aim of the study is to investigate progression in muscle affection in patients with pathogenic variants in the anoctamin 5 gene to:

1. investigate possible progression of disease over time
2. investigate good and reliable outcome measures

ELIGIBILITY:
Inclusion Criteria:

* Pathogenic variant in the anoctamin 5 gene
* Age more than 18 years

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathogenic variants in the anoctamin 5 gene are recruited from the Copenhagen Neuromuscular Center, Rigshospitalet, in Denmark.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in fat fraction during 3 years | 40 minutes
  Change in fat fraction (%) during 3 years in muscles from the whole body measured from Dixon MRI.

SECONDARY OUTCOMES:
Change in fatigue during 3 years | 5 minutes
  Change in fatigue during 3 years measured through the questionnaire 'fatigue severity score', FSS. 9 questions scoring from 1-7 where 7 correlates to "strongly agree". Higher score means more fatigue.
Change in quality of life during 3 years | 15 minutes
  Change in quality of life during 3 years measured through the questionnaire SF36. 36 questions. Higher score means higher quality of life.
Change in pain and function during 3 years | 10 minutes
  Change in pain and function in lower limbs during 3 years measured through the questionnaire 'low back pain rating scale ', LBPRS. 6 questions rated from 0-10 with 0 meaning no pain. Higher score means more pain.
Change in motor function during 3 years | 30 minutes
  Change in motor function during 3 years measured using the test the Motor Function Measure 32. 32 tasks to do, each task score 0-3. Higher score means better motor function.
Change in handgrip during 3 years | 10 minutes
  Change in handgrip during 3 years measured using a handgrip dynamometer.
Change in whole body muscle strenght during 3 years | 30 minutes
  Change in muscle strenght in whole body during 3 years measured using the technique 'manual muscle testning (MMT)' and the 'manual rating scale (MRC) '
Change in muscle strenght during 3 years | 30 minutes
  Change in muscle strenght in knee, hip and back during 3 years measured using a staionary dynamometer (a biodex dynamometer)
Change in balance during 3 years | 20 minutes
  Change in balance during 3 years measured using a biosway

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Neuromuscular Center, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided